CLINICAL TRIAL: NCT06548074
Title: Multicenter Pilot Project to Test the Healthy Parents and Children Enhancement (H-PACE) Program
Brief Title: H-PACE Program for the Improvement of Lifestyle Behaviors Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New Mexico State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1124059; NCI-2024-05449 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U54CA132381 (NIH); FHIRB0020386 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-07-26; First posted 2024-08-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Obesity
Keywords: physical activity (exercise); sedentary activity; sleep; fruit; vegetable
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Behavior Therapy; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (H-PACE program) (Experimental): See Detailed Description.
  Interventions: Behavioral: H-PACE Behavioral Intervention; Other: Accelerometer; Other: Questionnaire Administration; Other: Supportive Care

INTERVENTIONS:
Behavioral: H-PACE Behavioral Intervention — Participate in the H-PACE program
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Accelerometer — Wear an accelerometer
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Parents may participate in an optional virtual peer support group
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This clinical trial tests the effectiveness of a Healthy Parents and Children Enhancement (H-PACE) program for improving lifestyle behaviors among children. Proper nutrition and physical activity (PA) are essential parts of overall health. Together, they can decrease the risk of developing obesity as well as related diseases such as diabetes, heart disease, stroke, and several types of cancer. To address the prevalence of obesity and related diseases, programs focusing on increasing opportunities for active living and healthy eating are necessary. Multi-component school-based obesity prevention programs have demonstrated increases in PA and improvement in dietary habits; however, most afterschool programs are short term; evidence is needed to confirm long-term effects. Moreover, programs that involve parents have shown to be more successful in helping children choose healthier behaviors. Unfortunately, due to technological advancement, opportunities for children to be active in schools have become more limited in modern society. H-PACE program is based on the national childhood obesity prevention campaign designed to help families, schools, communities, and physicians to raise awareness of nutritional and PA daily guidelines. The H-PACE will encourage daily lifestyle behaviors (five or more servings of fruits and vegetables, two hours or less of recreational screen time, one hour of PA, zero sugary drinks, ten hours of sleep) that impact childhood obesity. This trial is being done to determine whether participating in the H-PACE program may help improve lifestyle behaviors among children.

DETAILED DESCRIPTION:
OUTLINE:

Children attend the H-PACE program comprising educational lessons over 30 minutes, PA over 30 minutes, and healthy snacks twice a week (BIW) for 12 weeks. The educational component includes 30-minute lessons on PA, fruits and vegetables, and sleep, followed by fun and entertaining games and activities. The PA component (30-minutes) comprises a variety of enjoyable activities including warm-up, main activities (e.g., walk/run/jog and aerobic fun games), and cool-down. The snack component introduces children to tasty and healthy foods and teaches children the skills to enable them to select and prepare healthy snack foods at school and at home. Snack education lessons emphasize the benefits of fruit and vegetable intake, and include a discussion of food composition (e.g., fat content, sugar, sodium). Children prepare healthy snack foods at home with parents once a week (QW) by taking home fruit and vegetable boxes with recipes for family-based engaging activities. Children also wear an accelerometer to monitor activity for 7 days at baseline and during week 11-12. Parents may participate in an optional virtual peer support group on study.

ELIGIBILITY:
Inclusion Criteria:

* Children in 3rd - 5th grade, 8-11 years of age, attending the afterschool program at the selected elementary schools.
* Parents/Guardians of the eligible child, who are ≥ 18 years old.
* Fluency in English or Spanish.

Exclusion Criteria:

* Children who are not in 3rd - 5th grade.
* Children not attending the afterschool program at the selected elementary schools.
* Parents/Guardians of the eligible child, who are < 18 years old.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage of children who attended more than 75% of program sessions (Feasibility) | Up to week 14
  Will be assessed using descriptive statistics. Will be considered a success from a feasibility standpoint if > 75% of participants meet the metric.
Percentage of children who completed more than 80% of assessment activities (Feasibility) | Up to week 14
  Will be assessed using descriptive statistics. Will be considered a success from a feasibility standpoint if > 75% of participants meet the metric.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Mendoza, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Dejan Magoc, PhD, Principal Investigator — New Mexico State University
Locations (2):
- United States (2):
  - New Mexico State University, Las Cruces, New Mexico
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT06548074/ICF_000.pdf